CLINICAL TRIAL: NCT06591507
Title: Perioperative Rehabilitation Therapy in Patients Undergoing Liver Transplantation: a Clinical Multicenter Study
Brief Title: Perioperative Rehabilitation Therapy in Patients Undergoing Liver Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT2024-ZJU-RCT1
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Liver Transplantation; Sarcopenia
Keywords: Liver transplantation; Sarcopenia; Branched-chain amino acids; Muscle rehabilitation
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Preoperative and Postoperative BCAA Nutritional Intervention (Experimental)
  Interventions: Dietary Supplement: BCAA Nutritional Intervention
- Preoperative and Postoperative BCAA Nutritional Intervention + Postoperative Muscle Rehabilitation (Experimental)
  Interventions: Dietary Supplement: BCAA Nutritional Intervention; Behavioral: Muscle Rehabilitation Training
- Postoperative BCAA Nutritional Intervention (Experimental)
  Interventions: Dietary Supplement: BCAA Nutritional Intervention
- Postoperative Muscle Rehabilitation (Experimental)
  Interventions: Behavioral: Muscle Rehabilitation Training
- Standard Nutritional Therapy (Placebo Comparator)
  Interventions: Dietary Supplement: Standard Nutritional Therapy

INTERVENTIONS:
Dietary Supplement: BCAA Nutritional Intervention — Patients will receive BCAA nutritional supplements. The supplement is taken orally twice daily, with each sachet containing 10g of powder, of which 6g is BCAA, and the remainder consists of preservatives and fruit flavorings to enhance palatability. The morning dose is taken with breakfast, and the second dose is taken as a late evening snack after dinner. For critically ill patients, enteral nutrition is provided instead. During each follow-up visit, patients are required to retain and submit all empty and unused sachets to accurately assess compliance. Dietitians will adjust the type and amount of food for each patient according to the guidelines of the European Society for Parenteral and Enteral Nutrition to ensure a total caloric intake of 35-40 kcal/kg and a protein intake of 1.2-1.5 g/kg (including BCAA supplements).
  Arms: Postoperative BCAA Nutritional Intervention; Preoperative and Postoperative BCAA Nutritional Intervention; Preoperative and Postoperative BCAA Nutritional Intervention + Postoperative Muscle Rehabilitation
Behavioral: Muscle Rehabilitation Training — Phase 1: Resistance Training (During Hospital Stay, First Month) Phase 2: Resistance Training (Home-Based, From Hospital Discharge Until 3 Months Post-Surgery) Phase 3: Physical Activity Training (Post-Surgery, After 3 Months)
  Arms: Postoperative Muscle Rehabilitation; Preoperative and Postoperative BCAA Nutritional Intervention + Postoperative Muscle Rehabilitation
Dietary Supplement: Standard Nutritional Therapy — Standard Nutritional Therapy
  Arms: Standard Nutritional Therapy

SUMMARY:
Patients undergoing liver transplantation frequently experience a reduction in skeletal muscle mass, malnutrition, and decreased levels of physical activity. These complications can adversely affect early postoperative recovery and the therapeutic effect of the transplant. This clinical study aims to investigate the effects of nutritional supplementation and rehabilitation therapy on sarcopenia associated with liver transplantation in adults. The goal is to establish a comprehensive perioperative intervention strategy to reduce the incidence of postoperative sarcopenia and improve transplantation outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Patients with end-stage liver disease who meet the criteria for liver transplantation (for liver cancer cases, only recipients meeting specific standards are included).
3. Complete clinical information, including documented pre-transplant muscle status (e.g., preoperative CT scans and handgrip strength tests).
4. High compliance with treatment, fully capable of independent action or having at least one assistant.
5. No contraindications to the planned interventions.

Exclusion Criteria:

1. Presence of musculoskeletal disorders before transplantation, such as myositis, idiopathic muscle atrophy, or history of hip surgery within the past three months.
2. Coexisting severe cardiovascular or cerebrovascular diseases, infectious diseases, or epilepsy.
3. Liver transplantation due to autoimmune liver disease or drug-induced liver failure.
4. Re-transplantation, multi-organ transplantation, living donor liver transplantation, split liver transplantation, or pediatric liver transplantation.
5. ABO-incompatible liver transplantation.
6. Incomplete clinical information.
7. Difficulty in follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival | From enrollment to the end of follow-up at 2 years
  At the 2-year mark, record the survival status of each patient (alive or deceased).

SECONDARY OUTCOMES:
Muscle mass | From enrollment to the end of treatment at 6 months
  Muscle mass can be assessed using various methods, including CT-based Skeletal Muscle Index (SMI) calculation at the L3 vertebra, which measures the cross-sectional area of muscle normalized by height; handgrip strength testing, which evaluates muscle function; bioelectrical impedance analysis (BIA) for body composition; MRI for precise muscle volume measurements; and dual-energy X-ray absorptiometry (DXA) for assessing lean body mass. These methods provide a comprehensive evaluation of muscle health.

IPD SHARING:
Plan to Share IPD: Undecided